CLINICAL TRIAL: NCT07005648
Title: Population-based Cross-sectional Observational Study for a Brazilian Registry of Menopausal Women and Associated Factors Related to Clinical Profile, Socioeconomic Aspects, Social Disparities, Access to Healthcare, Quality of Life, and Knowledge About Menopause
Brief Title: Brazilian Registry of Menopausal Health
Status: Not yet recruiting | Type: Observational
Sponsor: Science Valley Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RENEW
Record Dates: First submitted 2025-04-24; First posted 2025-06-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Menopause
Keywords: Menopause; Post Menopause; Menopause Transition; Climateric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 617 participants = 35 to 44 years old
- 509 participants = 45 to 54 years old
- 466 participants = 55 to 65 years old

SUMMARY:
The Brazilian Registry of Menopausal Health is a national study aimed to better understand the health and quality of life of participants aged 35 to 65 who are in the menopausal transition or postmenopausal phase, including cisgender women and transgender men.The study's hypothesis is that significant regional and socioeconomic disparities influence individuals' health, knowledge, and perception of menopause.

DETAILED DESCRIPTION:
The Brazilian Registry of Menopausal Health, called RENEW (Registry of ENdocrine Changes in midlifE Women), is an observational, cross-sectional, population-based study conducted with the objective of characterizing the epidemiological aspects of the Brazilian population during the menopausal transition and postmenopause, as well as the factors associated with clinical profiles and symptomatology, socioeconomic conditions, social inequalities, access to healthcare services, quality of life, and knowledge about menopause.

The study will include cisgender women and transgender men who have not undergone surgical or hormonal gender reassignment of secondary sexual characteristics, aged between 35 and 65 years, who seek outpatient care in public or private healthcare services.

A total of 1,592 participants will be enrolled, with 617, 509, and 466 participants in the respective age groups of 35-44, 45-54, and 55-65 years, proportionally stratified across the 27 state capitals of Brazil. These age groups will be used solely for the purpose of sample stratification.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 35 and 65 years attending medical consultation at public and private outpatient health services;
2. Ability to confirm voluntary participation and sign the Informed Consent Form

Exclusion Criteria:

1. Inability to respond to the interview for any reason
2. Suspected or confirmed pregnancy
3. Lactation
4. Uncontrolled diabetes
5. Uncontrolled arterial hypertension
6. Uncontrolled thyroid disorders
7. Grade 3 obesity, defined by a BMI equal to or greater than 40.0 kg/m²
8. Diagnosis of psychiatric disorders that may compromise participation in the interview
9. Previous hysterectomy
10. Previous oophorectomy
11. Current use of illicit drugs

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women or transgender men who have not undergone surgical or hormonal reassignment of secondary sexual characteristics.
Study Population: Cisgender women or transgender men who have not undergone surgical or hormonal reassignment of secondary sexual characteristics, aged between 35 and 65 years, seeking outpatient care in public or private healthcare services.
Sampling Method: Non-Probability Sample
Enrollment: 1592 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants aged 35 to 65 classified as being in the menopausal transition or postmenopause. | Day 1 (during the medical appointment)
  Definition of menopausal status. Premenopause: regular menstrual cycles, corresponding to the reproductive period preceding menopause; Menopausal transition: characterized by irregular menstrual cycles and amenorrhea for less than 12 months.
  Postmenopause: amenorrhea for more than 12 months.

SECONDARY OUTCOMES:
Proportion of participants in each menopausal status. | Day 1 (during the medical appointment)
  Premenopause; Menopausal transition; Postmenopause.
Characterization of the clinical profile. | Day 1 (during the medical appointment)
  This outcome measure includes a structured assessment of variables related to the participant's gynecologic and clinical history: age at menarche, menstruation status, date of last menstruation, age at last menstruation, personal medical history, and comorbidities.
  These variables and the summary statistics (when applicable) will be aggregated to produce a standardized clinical profile report for each participant.
Characterization of knowledge and self-perception of menopause. | Day 1 (during the medical appointment)
  This outcome measure includes a structured assessment of participants' understanding and personal perspective regarding menopause. The evaluation comprises the following elements: perception of menopause, definitions of menopause, history of hormone therapy (HT) use, perception and expectations regarding HT, and perceived impact of HT on menopause experience.
  These variables will be aggregated to generate a descriptive profile of knowledge and self-perception of menopause for each participant.
Characterization of the anthropometric and physiological profile. | Day 1 (during the medical appointment)
  This outcome measure includes anthropometric and physiological parameters: weight (in kilograms), height (in centimeters), body mass index (BMI, calculated as weight/height² in kg/m²), waist circumference (in centimeters), hip circumference (in centimeters), and blood pressure (in mmHg). These variables will be aggregated to generate an anthropometric profile for each participant, allowing for descriptive and comparative analysis of body composition and cardiovascular markers.
Characterization of General Health Profile. | Day 1 (during the medical appointment)
  This outcome measure includes a structured assessment of the participant's self-reported health status and medical history. It comprises self-perception of health, history of surgeries, pre-existing comorbidities, and current use of medications.
  These variables will be aggregated into a descriptive health profile for each participant.
Characterization of Laboratory Profile. | Day 1 (during the medical appointment)
  This outcome measure includes laboratory test results related to metabolic, hormonal, and glycemic profiles. The following biomarkers will be collected: Thyroid-Stimulating Hormone (TSH), Free Thyroxine (T4), Luteinizing Hormone (LH), Follicle-Stimulating Hormone (FSH), Estradiol, Progesterone, Total Cholesterol, Low-Density Lipoprotein Cholesterol (LDL), High-Density Lipoprotein Cholesterol (HDL), Triglycerides, Fasting Glucose, and Glycated Hemoglobin. These results will be aggregated to form a laboratory profile for each participant.
Characterization of the social profile. | Day 1 (during the medical appointment)
  This outcome measure includes a structured assessment of socioeconomic profile, access to healthcare and employment status. The variables assessed in socioeconomic classification are according to the Brazilian Association of Companies and Research (ABEP) and were used to analyze the socioeconomic level, which includes the educational level of the head of household, and includes questions about family income, possession of public items and services offered in its residence. These data will be aggregated to generate a social profile for each participant.
Characterization of the demographic profile. | Day 1 (during the medical appointment)
  This outcome measure includes key demographic variables relevant to reproductive and social background: marital status, education level, race/skin color, number of children, number of pregnancies, and number of abortions. These data will be aggregated to produce a comprehensive understanding of the demographic participant profile.
Characterization of lifestyle profile. | Day 1 (during the medical appointment)
  This outcome measure includes a structured assessment of lifestyle-related behaviors. The variables assessed are history of smoking, physical activity practice, alcohol consumption, and use of psychoactive substances. These variables will be aggregated to produce a lifestyle profile for each participant.
Total score and quantitative domains of the QSM/WHQ questionnaire [Women's Health Questionnaire (WHQ) / Questionário da Saúde da Mulher (QSM); applicable to women aged 45 to 65 years]. | Day 1 (during the medical appointment)
  Women's health questionnaire (WHQ/QSM) is used to evaluate quality of life. This validated 36-item questionnaire measures changes in nine domains of physical and emotional health associated with the menopause transition. Analysis results in a score between 0.00 and 1.00, where higher scores are associated with worse symptomology and quality of life. A change of 0.10-0.20 is clinically meaningful.
Total score and quantitative domains of the SF-36 questionnaire [36-Item Short-Form Health Survey]. | Day 1 (during the medical appointment)
  The SF-36 is a 36-item, 8-domain questionnaire used to assess overall health: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health
Total score and quantitative domains of the WPAI-GH questionnaire [WPAI-GH (Work Productivity and Activity Impairment - General Health)]. | Day 1 (during the medical appointment)
  The WPAI (Work Productivity and Activity Impairment) is questionnaire created as a patient-reported quantitative assessment. This questionnaire has 6 questions, which are used to calculate 4 types of scores; which are absenteeism (work time missed), presenteeism (reduced on the job effectiveness), work productivity loss (overall work impairment) and activity impairment. The scores are expressed in percentage with higher numbers indicating greater impairment and less productivity
Classification of anxiety according to the GAD-7 questionnaire [Generalized Anxiety Disorder scale]. | Day 1 (during the medical appointment)
  The GAD-7 is a self-administered questionnaire that assesses generalized anxiety, composed of seven questions covering aspects such as excessive worry, difficulty controlling worry, irritability, muscle tension, fatigue, difficulty relaxing, and sleep problems. Each question is scored from 0 to 3, with a severity score ranging from 0 to 21. Cutoff points are ≥5 for mild anxiety, ≥10 for moderate anxiety, and ≥15 for severe anxiety.
Classification of depression according to the PHQ-9 questionnaire [Patient Health Questionnaire-9 (PHQ-9)]. | Day 1 (during the medical appointment)
  The PHQ-9 is a self-administered questionnaire focused on depression, consisting of nine questions addressing aspects like diminished interest, depressed mood, fatigue, sleep issues, appetite changes, low self-esteem, difficulty concentrating, slowed movements or agitation, and suicidal thoughts. Each question is scored from 0 to 3, with a severity score from 0 to 27. Severe depression is indicated by a score >16.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiane B de Souza, MD, Principal Investigator — Science Valley Research Institute
Locations (1):
- Centro de Pesquisa Unidade Morumbi - Science Valley Research Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thurston RC, Joffe H. Vasomotor symptoms and menopause: findings from the Study of Women's Health across the Nation. Obstet Gynecol Clin North Am. 2011 Sep;38(3):489-501. doi: 10.1016/j.ogc.2011.05.006. PMID 21961716
- [Background] Flores VA, Pal L, Manson JE. Hormone Therapy in Menopause: Concepts, Controversies, and Approach to Treatment. Endocr Rev. 2021 Nov 16;42(6):720-752. doi: 10.1210/endrev/bnab011. PMID 33858012
- [Background] Mehta J, Kling JM, Manson JE. Risks, Benefits, and Treatment Modalities of Menopausal Hormone Therapy: Current Concepts. Front Endocrinol (Lausanne). 2021 Mar 26;12:564781. doi: 10.3389/fendo.2021.564781. eCollection 2021. PMID 33841322
- [Background] Davis SR, Taylor S, Hemachandra C, Magraith K, Ebeling PR, Jane F, Islam RM. The 2023 Practitioner's Toolkit for Managing Menopause. Climacteric. 2023 Dec;26(6):517-536. doi: 10.1080/13697137.2023.2258783. Epub 2023 Dec 1. PMID 37902335
- [Background] Oliveira GMM, Almeida MCC, Arcelus CMA, Neto Espindola L, Rivera MAM, Silva-Filho ALD, Marques-Santos C, Fernandes CE, Albuquerque CJDM, Freire CMV, Izar MCO, Costa MENC, Castro ML, Lemke VMG, Lucena AJG, Brandao AA, Macedo AVS, Polanczyk CA, Lantieri CJB, Nahas EP, Alexandre ERG, Campana EMG, Braganca EOV, Colombo FMC, Barbosa ICQ, Rivera IR, Kulak J, Moura LAZ, Pompei LM, Baccaro LFC, Barbosa MM, Rodrigues MAH, Albernaz MA, Decoud MSP, Paiva MSMO, Sanchez-Zambrano MB, Campos MDSB, Acevedo M, Ramirez MS, Souza OF, Medeiros OO, Carvalho RCM, Machado RB, Silva SCTFD, Rodrigues TCV, Avila WS, Costa-Paiva LHSD, Wender MCO. Brazilian Guideline on Menopausal Cardiovascular Health - 2024. Arq Bras Cardiol. 2024 Aug 16;121(7):e20240478. doi: 10.36660/abc.20240478. No abstract available. English, Portuguese. PMID 39166619
- [Background] Duralde ER, Sobel TH, Manson JE. Management of perimenopausal and menopausal symptoms. BMJ. 2023 Aug 8;382:e072612. doi: 10.1136/bmj-2022-072612. PMID 37553173